CLINICAL TRIAL: NCT04344483
Title: Effect of Lidocaine and Adrenaline Soaked Gauze Versus Normal Saline Soaked at Skin Graft Donor Site of Thigh: A Randomized Control Trial
Brief Title: Effect of Lidocaine and Adrenaline Soaked Gauze Versus Normal Saline Soaked at Skin Graft Donor Site of Thigh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Zaara Zahid, Principle investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1506
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Non-healing Wound
MeSH Terms: interventions — Lidocaine; Epinephrine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Patients with non healing wound who will otherwise be healthy will be recruited in the study and will randomly assign groups. One group will receive Adrenaline and Lidocaine soaked gauze and the second group will be a control group who will receive normal saline soaked gauze.
Who Masked: Participant
Masking Description: Patients will be recruited in the study by closed envelope technique and the study will be single blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A ( Lidocaine + Adrenaline) (Active Comparator): Group A patients will receive 2% Lidocaine and 1:100,000 adrenaline soaked gauze over skin graft donor site of thigh per operatively for 10 minutes. After 10 minutes this dressing will be removed and sufratul dressing will be applied over donor site.
  Interventions: Drug: 2% Lidocaine and 1:100,000 Adrenaline
- Group B ( Normal Saline) (Placebo Comparator): Group B patients will receive normal saline soaked gauze over skin graft donor site of thigh intraoperatively for 10 minutes. After 10 minutes this dressing will be removed and sufratul dressing will be applied over donor site
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: 2% Lidocaine and 1:100,000 Adrenaline — Topical application of 2% Lidocaine and 1:100,000 Adrenaline in the form of dressing will be applied over skin graft donor site of thigh for 10 minutes.
  Arms: Group A ( Lidocaine + Adrenaline)
Drug: Normal saline — Topical application of Normal saline will be applied over skin graft donor site of thigh as a control group.
  Arms: Group B ( Normal Saline)

SUMMARY:
Investigator is studying the effects of Lidocaine and Adrenaline Soaked Gauze vs Normal Saline Soaked Gauze at Skin Graft Donor Site of Thigh.

Haemostatic effect, epithelization and post operative pain will be assessed on follow up.

DETAILED DESCRIPTION:
After admission participants will be randomized either to be in Group A or Group B. Closed envelop technique will be used for random assignment of the patients.

Group A will be receiving 2% lidocaine and 1:100,000 adrenaline soaked gauze while group B will be given only normal saline soaked gauze at donor-site for ten minutes.

The primary end point of study is intraoperative bleeding. The secondary end points of study include no. of dressings required in first 24 hours after surgery, donor site epithelization at 14th post-operative day, post-operative pain in first 24 hours after surgery along with systemic analgesia requirement after surgery.

ELIGIBILITY:
Inclusion Criteria:

* • Patients of both the gender of age > 15 years

  * Multiple donor-sites

Exclusion Criteria:

Bleeding disorder

* Concomitant injuries
* Donor site other than thigh
* Previously harvested donor-site
* Patients on antiplatelet medications

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Intra operatieve bleeding | per operative
  Intra-operative Bleeding from donor site of graft will be assessed per operatively as being normal or more than normal.
Post operative bleeding | 24 hours
  post operative bleeding will be assesd in post operative period by number of dressings required.
Post operative pain | 24 hours
  post operative pain will be assessed in the post operative period by visual analog score. Score ranges from 0 to 10 with 0 indicating no pain whereas 10 is worst pain.
Analgesia requirement | 24 hours
  Post operative analgesia requirement of patient will be observed by number of medications required

SECONDARY OUTCOMES:
Epithelization of donor site | 14 days
  Epithelization over donor site will be assessed on 14th post operative day by subjective assesment

CONTACTS AND LOCATIONS:
Locations (1):
- Zaara Zahid, Karachi, Sindh, Pakistan

REFERENCES:
- [Result] Gacto P, Miralles F, Pereyra JJ, Perez A, Martinez E. Haemostatic effects of adrenaline-lidocaine subcutaneous infiltration at donor sites. Burns. 2009 May;35(3):343-7. doi: 10.1016/j.burns.2008.06.019. Epub 2008 Oct 23. PMID 18950945
- See also: Gacto P, Miralles F, Pereyra J, Perez A, Martinez E. Haemostatic effects of adrenaline-lidocaine subcutaneous infiltration at donor sites. Burns. 2009;35(3):343-7. — https://www.ncbi.nlm.nih.gov/pubmed/18950945